CLINICAL TRIAL: NCT02263911
Title: Relative Bioavailability of the Baricitinib (LY3009104) Commercial Tablet Compared to the Phase 2 Tablets and the Effect of Food on the Bioavailability of the Commercial Tablet in Healthy Japanese Subjects
Brief Title: A Study of Baricitinib in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14612; I4V-MC-JAGO (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Baricitinib Test Treatment 1 (T1) (Experimental): Single oral dose of 2 × 4 milligram (mg) baricitinib commercial formulation tablet fasted on Day 1 in one of five periods.
  Interventions: Drug: Baricitinib
- Baricitinib Reference Treatment 1 (R1) (Experimental): Single oral dose of 1 × 8 mg baricitinib Phase 2 tablet fasted on Day 1 in one of five periods.
  Interventions: Drug: Baricitinib
- Baricitinib Test Treatment 2 (T2) (Experimental): Single oral dose of 1 × 4 mg baricitinib commercial formulation tablet fasted on Day 1 in one of five periods.
  Interventions: Drug: Baricitinib
- Baricitinib Reference Treatment 2 (R2) (Experimental): Single oral dose of 1 × 4 mg baricitinib Phase 2 tablet fasted on Day 1 in one of five periods.
  Interventions: Drug: Baricitinib
- Baricitinib Test Treatment 2 with Meal (T2F) (Experimental): Single oral dose of 1 × 4 mg baricitinib commercial formulation tablet after food intake on Day 1 in one of five periods.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104

SUMMARY:
The purpose of this study is to understand the relationship of 3 different dosage forms of baricitinib. This study will also explore the effect of food on how the body absorbs baricitinib. This study will last about 5 weeks, not including screening. Screening is required within 28 days prior to the date of first dosing.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy Japanese male and female (women not of child-bearing potential or after menopause), as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.5 to 29.9 kilogram per square meter (kg/m^2)
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure as determined by the investigator
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Are women who are pregnant or lactating
* Have used or intend to use over-the-counter or prescription medication, including herbal medications, within 14 days prior to dosing and during the study.
* Have donated blood of more than 400 milliliter (mL) in the last 12 weeks (males) or in the last 16 weeks (females), or any blood donation (including apheresis) within the last 4 weeks, or total volume of blood donation within 12 months is 1200 mL (males) or 800 mL (females) at screening.
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to abide by alcohol restrictions
* Are participants who currently smoke more than 10 cigarettes per day (or equivalent in tobacco or nicotine products) or are unwilling to abide by smoking restrictions
* Have a current or recent history of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have an absolute neutrophil count (ANC) less than 2000 cells/microliter (µL)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hachiōji, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Baricitinib Dosing Sequence 1: Single oral dose of study drug daily on 5 occasions: Test Treatment 1 (T1) = Baricitinib 2 × 4 milligram (mg) commercial formulation tablets in a fasted state, Reference Treatment 1 (R1) = Baricitinib 1 × 8 mg Phase 2 tablet in a fasted state, Test Treatment 2 (T2) = Baricitinib 1 × 4 mg commercial formulation tablet in a fasted state, Reference Treatment 2 (R2) = Baricitinib 1 × 4 mg Phase 2 tablet in a fasted state, and (T2F) = Baricitinib 2 × 4 mg commercial formulation tablets in a fed state. Dosing occasions were separated by at least 7 days.
- Baricitinib Dosing Sequence 2: Single oral dose of study drug daily on 5 occasions: R1 = Baricitinib 1 × 8 mg Phase 2 tablet in a fasted state, T1 = Baricitinib 2 × 4 mg commercial formulation tablets in a fasted state, R2 = Baricitinib 1 × 4 mg Phase 2 tablet in a fasted state, T2 = Baricitinib 1 × 4 mg commercial formulation tablet in a fasted state, and T2F = Baricitinib 2 × 4 mg commercial formulation tablets in a fed state. Dosing occasions were separated by at least 7 days.
- Baricitinib Dosing Sequence 3: Single oral dose of study drug daily on 5 occasions: T1 = Baricitinib 2 × 4 mg commercial formulation tablets in a fasted state, R1 = Baricitinib 1 × 8 mg Phase 2 tablet in a fasted state, R2 = Baricitinib 1 × 4 mg Phase 2 tablet in a fasted state, T2 = Baricitinib 1 × 4 mg commercial formulation tablet in a fasted state, and T2F = Baricitinib 2 × 4 mg commercial formulation tablets in a fed state. Dosing occasions were separated by at least 7 days.
- Baricitinib Dosing Sequence 4: Single oral dose of study drug daily on 5 occasions: R1 = Baricitinib 1 × 8 mg Phase 2 tablet in a fasted state, T1 = Baricitinib 2 × 4 mg commercial formulation tablets in a fasted state, T2 = Baricitinib 1 × 4 mg commercial formulation tablet in a fasted state, R2 = Baricitinib 1 × 4 mg Phase 2 tablet in a fasted state, and T2F = Baricitinib 2 × 4 mg commercial formulation tablets in a fed state. Dosing occasions were separated by at least 7 days.
Period: Period 1
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 1 Washout
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 Washout
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 Washout
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 Washout
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Baricitinib Dosing Sequence 1 | Baricitinib Dosing Sequence 2 | Baricitinib Dosing Sequence 3 | Baricitinib Dosing Sequence 4
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All randomized participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Baricitinib
Time Frame: Day 1: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, and 48 Hours Post-dose
Population: All randomized participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Baricitinib T1: Baricitinib 2 × 4 mg commercial formulation tablets given orally (PO) once daily (QD) in the fasted state on Day 1 in one of five periods.
- Baricitinib R1: Baricitinib 1 × 8 mg Phase 2 tablet administered PO QD in the fasted state on Day 1 in one of five periods.
- Baricitinib T2: Baricitinib 1 × 4 mg commercial formulation tablet administered PO QD in the fasted state on Day 1 in one of five periods.
- Baricitinib R2: Baricitinib 1 × 4 mg Phase 2 tablet administered PO QD in the fasted state on Day 1 in one of five periods.
- Baricitinib T2F: Baricitinib 1 × 4 mg commercial formulation tablet administered PO QD with a low-fat meal on Day 1 in one of five periods.
Arm/Group | Baricitinib T1 | Baricitinib R1 | Baricitinib T2 | Baricitinib R2 | Baricitinib T2F
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nanogram*hour/milliliter (ng*h/mL) | 626 (19) | 584 (20) | 297 (17) | 301 (17) | 254 (14)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Last Measurable Concentration (AUC[0-tlast]) of Baricitinib
Time Frame: Day 1: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, and 48 Hours Post-dose
Population: All randomized participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Baricitinib T1: Baricitinib 2 × 4 mg commercial formulation tablets administered PO QD in the fasted state on Day 1 in one of five periods.
Arm/Group | Baricitinib T1 | Baricitinib R1 | Baricitinib T2 | Baricitinib R2 | Baricitinib T2F
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng*h/mL | 622 (19) | 580 (20) | 294 (17) | 298 (17) | 251 (14)

3. Primary Outcome: PK: Maximum Concentration (Cmax) of Baricitinib
Time Frame: Day 1: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36, and 48 Hours Post-dose
Population: All randomized participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Baricitinib T1: Baricitinib 2 × 4 mg commercial formulation tablet administered PO QD in the fasted state on Day 1 in one of five periods.
Arm/Group | Baricitinib T1 | Baricitinib R1 | Baricitinib T2 | Baricitinib R2 | Baricitinib T2F
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nanogram/milliliter (ng/mL) | 107 (29) | 103 (27) | 50.7 (25) | 53.1 (18) | 45.1 (31)

ADVERSE EVENTS:
Arm/Group | Baricitinib T1 | Baricitinib R1 | Baricitinib T2 | Baricitinib R2 | Baricitinib T2F
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days